CLINICAL TRIAL: NCT05378971
Title: Clinical Research of Pomalidomide Maintenance Therapy for Primary Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Collaborators: Beijing Health Alliance Charitable Foundation (Unknown)
Responsible Party: Principal Investigator, Hao Zhang, Master, associate chief physician, Principal Investigator, LanZhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POMLDYY
Record Dates: First submitted 2022-04-21; First posted 2022-05-18 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Maintenance treatment; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Intervention Model Description: Patients enrolled were divided into two categories: 1) patients suitable for Autologous Hematopoietic Stem Cell Transplantation(ASCT) started pomalidomide maintenance therapy 3 months after ASCT; 2) patients not suitable for ASCT started pomalidomide maintenance therapy after induction and consolidation therapy to achieve maximum efficacy. Dosing on days 1-21, 2 mg daily for 28 days as a cycle, for a total duration of 36 months or the onset of disease progression, intolerable adverse events.
Masking Description: Subjects and researchers can know which treatment is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Primary MM patients started maintenance therapy after 3 months of ASCT or after maximum efficacy was achieved with induction and consolidation therapy. All patients will receive pomalidomide 1 mg daily on days 1 through 21 of each 28-day cycle.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide, 2mg/d, d1-21; treatment cycles every 28days
  Other Names: Pomalyst

SUMMARY:
The trial is a single-center, single-arm, prospective clinical study with a planned enrollment of 15 patients with primary Multiple myeloma(MM), aiming to investigate the efficacy and safety of maintenance therapy with Pomalidomide in patients with primary MM. Patients enrolled were divided into two categories: 1) patients suitable for Autologous Hematopoietic Stem Cell Transplantation(ASCT) started pomalidomide maintenance therapy 3 months after ASCT; 2) patients not suitable for ASCT started pomalidomide maintenance therapy after induction and consolidation therapy to achieve maximum efficacy. Dosing on days 1-21, 2 mg daily for 28 days as a cycle, for a total duration of 36 months or the onset of disease progression, intolerable adverse events. 2-year progression-free survival (2y-PFS) was used as the primary study endpoint, 2-year overall survival (2y-OS), complete remission rate (CR), very good partial remission rate (VGPR), and negative rate of minimal residual disease(MRD) were secondary study endpoints, and the incidence of adverse events (AEs) was assessed.

DETAILED DESCRIPTION:
Maintenance regimens based on thalidomide and lenalidomide have been shown in numerous clinical trials to significantly improve PFS in patients, but the use of thalidomide is limited by adverse effects such as peripheral neurotoxicity and post-relapse drug resistance. Pomalidomide is a third-generation immunomodulator with a similar structure to thalidomide and lenalidomide, but with stronger anti-MM activity and a similar safety profile. The known mechanisms of action include (1) immunomodulatory effects (2) direct antitumor effects (3) anti-angiogenic activity. (4) Effects on the bone marrow microenvironment. The most common toxicities of pomalidomide include bone marrow suppression, skin reactions, gastrointestinal reactions, and infections, etc. Peripheral neuropathy is less common than thalidomide, and the incidence of thromboembolism is <5%. Pomalidomide is currently used mainly in the treatment of relapsed refractory adult MM, and exploration in post-ASCT maintenance therapy is currently ongoing (NCT01745588). Several retrospective analyses suggest that low-dose pomalidomide may have potential in the maintenance treatment of patients with MM. Therefore, investigators developed a maintenance regimen of low-dose pomalidomide to assess the value of maintenance therapy in MM patients who underwent ASCT or who were not suitable for ASCT. Such regimens may reduce drug toxicity and provide greater clinical benefit for patients with MM.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed as initially diagnosed with symptomatic MM by the diagnostic criteria of International Myeloma Working Group(IMWG), aged ≥ 18 years.
2. Subject undergoing ASCT who have had prior induction therapy for no more than 12 months and whose disease has not progressed within 3 months of ASCT.
3. Subject who are not candidates for ASCT have reached maximum efficacy after induction and consolidation therapy.
4. Eastern Cooperative Oncology Group (ECOG) physical status score of 0-3.
5. Serum transaminase levels less than three times the upper limit of normal, serum total bilirubin levels not exceeding 35 umol/L, serum creatinine levels less than 177 umol/L, absolute neutrophil values greater than 1.0 x 10^9/L, and platelet counts greater than 75 x 10^9/L.
6. Subject of childbearing potential must use two reliable methods of contraception simultaneously or have absolutely no sexual relations with the opposite sex for 4 weeks prior to initiation of treatment, during treatment, during suspension of dosing and for 4 weeks after termination of treatment, and women of childbearing potential agree to perform monthly pregnancy tests until 4 weeks after discontinuation of study drug.
7. Subject voluntarily enrolled in this study and signed an informed consent form.

Exclusion Criteria:

1. Subject has 17p-, 1q21 amplification, t(4;14), t(14;16), t(14;20), t(11;14), and p53 mutation.
2. Subject who, in the judgment of the investigator, cannot tolerate pomalidomide treatment or are allergic to lenalidomide or thalidomide drugs.
3. Subject with a diagnosis of nonsecretory MM (meaning subjects with completely nonsecretory MM or subjects with a small amount of free light chain but with less than 100 mg/L of affected light chain).
4. with central nervous system involvement.
5. subject with peripheral neuropathy ≥ grade 3.
6. subject with known active hepatitis B virus (HBV-DNA ≥ l × 103 copies/mL or HBV-DNA > 200 IU/mL) or hepatitis C virus (HCV), or serologically positive for human immunodeficiency virus (HIV).
7. Subject with concurrent other neoplasms or a prior history of neoplasms or antineoplastic therapy (including major surgery) within the last 4 weeks, except for the following neoplastic diseases or those who have lived tumor-free for ≥ 3 years to date: basal cell carcinoma of the skin, squamous epithelial cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histologic findings of prostate cancer (TNM clinical stage of T1a or T1b) or treated prostate cancer.
8. Subject with coexisting serious infectious disease.
9. Subject who refuse to use a reliable form of contraception during pregnancy and lactation or at an appropriate age.
10. Subject with active new thrombosis or unwilling to undergo antithrombotic therapy.
11. Subject who, in the opinion of the investigator, are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival(2y-PFS) | up to 24 months.
  2y-PFS was defined as the proportion of patients who reached at least 2 years from the first day of treatment to the time of disease progression or death.

SECONDARY OUTCOMES:
2-year overall survival(2y-OS) | up to 24 months.
  2y-OS was defined as the proportion of patients with a time from the first day of treatment to death of at least 2 years.
Complete remission(CR) | up to 24 months.
  It includes strict complete remission (sCR), CR: negative serum and urine immunofixation electrophoresis and bone marrow plasma cells <5%; sCR: normal serum free light chain ratio and absence of clonal plasma cells in bone marrow confirmed by immunohistochemistry on the basis of meeting CR criteria;
very good partial remission(VGPR) | up to 24 months.
  VGPR: undetectable M protein by serum protein electrophoresis but still positive by serum and and urine immunofixation electrophoresis, or ≥90% reduction in M protein and urine M protein <100 mg/24h.
negative rate of minimal residual disease | up to 24 months.
  Flow cytometry was used to detect cells with abnormal immunophenotype, and residual tumor cells <10-4 were considered negative.
adverse events | Adverse event reports are collected once a month during treatment, up to 24 months.
  number of participants with treatment-related adverse events as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhang, Principal Investigator — The First Hospital of Lanzhou University,Lanzhou, Gansu, China
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
After the completion of the clinical trial, we will choose whether to disclose the result according to the relevant regulations of the Chinese Genetic Office.

REFERENCES:
- [Background] Costa LJ, Brill IK, Omel J, Godby K, Kumar SK, Brown EE. Recent trends in multiple myeloma incidence and survival by age, race, and ethnicity in the United States. Blood Adv. 2017 Jan 4;1(4):282-287. doi: 10.1182/bloodadvances.2016002493. eCollection 2017 Jan 10. PMID 29296944
- [Background] Rawstron AC, Child JA, de Tute RM, Davies FE, Gregory WM, Bell SE, Szubert AJ, Navarro-Coy N, Drayson MT, Feyler S, Ross FM, Cook G, Jackson GH, Morgan GJ, Owen RG. Minimal residual disease assessed by multiparameter flow cytometry in multiple myeloma: impact on outcome in the Medical Research Council Myeloma IX Study. J Clin Oncol. 2013 Jul 10;31(20):2540-7. doi: 10.1200/JCO.2012.46.2119. Epub 2013 Jun 3. PMID 23733781
- [Background] Munshi NC, Avet-Loiseau H, Rawstron AC, Owen RG, Child JA, Thakurta A, Sherrington P, Samur MK, Georgieva A, Anderson KC, Gregory WM. Association of Minimal Residual Disease With Superior Survival Outcomes in Patients With Multiple Myeloma: A Meta-analysis. JAMA Oncol. 2017 Jan 1;3(1):28-35. doi: 10.1001/jamaoncol.2016.3160. PMID 27632282
- [Background] Liu H, McCarthy P. New developments in post-transplant maintenance treatment of multiple myeloma. Semin Oncol. 2013 Oct;40(5):602-9. doi: 10.1053/j.seminoncol.2013.07.008. PMID 24135405
- [Background] Rios-Tamayo R, Martin-Garcia A, Alarcon-Payer C, Sanchez-Rodriguez D, de la Guardia AMDVD, Garcia Collado CG, Jimenez Morales A, Jurado Chacon M, Cabeza Barrera J. Pomalidomide in the treatment of multiple myeloma: design, development and place in therapy. Drug Des Devel Ther. 2017 Aug 22;11:2399-2408. doi: 10.2147/DDDT.S115456. eCollection 2017. PMID 28860711
- [Background] Rychak E, Mendy D, Shi T, Ning Y, Leisten J, Lu L, Miller K, Narla RK, Orlowski RZ, Raymon HK, Bjorklund CC, Thakurta A, Gandhi AK, Cathers BE, Chopra R, Daniel TO, Lopez-Girona A. Pomalidomide in combination with dexamethasone results in synergistic anti-tumour responses in pre-clinical models of lenalidomide-resistant multiple myeloma. Br J Haematol. 2016 Mar;172(6):889-901. doi: 10.1111/bjh.13905. Epub 2016 Feb 23. PMID 26914976
- [Background] Richardson PG, Mark TM, Lacy MQ. Pomalidomide: new immunomodulatory agent with potent antiproliferative effects. Crit Rev Oncol Hematol. 2013 Oct;88 Suppl 1:S36-44. doi: 10.1016/j.critrevonc.2013.02.001. Epub 2013 Jun 17. PMID 23786844
- [Background] Atieh T, Hubben A, Faiman B, Valent J, Samaras CJ, Khouri J. Pomalidomide-based maintenance post-autologous hematopoietic cell transplantation in multiple myeloma: a case series. Ann Hematol. 2019 Oct;98(10):2457-2459. doi: 10.1007/s00277-019-03772-1. Epub 2019 Aug 7. No abstract available. PMID 31392460